CLINICAL TRIAL: NCT06867783
Title: EVALUATION OF EARLY FAMILY AND MULTIFAMILY INTERVENTION FOR YOUNG CHILDREN WITH AUTISM SPECTRUM DISORDERS
Brief Title: EVALUATION FOR YOUNG CHILDREN WITH AUTISM SPECTRUM DISORDERS
Acronym: coquille
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Pierre LECARPENTIER, MBBS, psychiatrist and investigator, Centre hospitalier de Ville-Evrard, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10477M-COQUILLE
Record Dates: First submitted 2025-01-07; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder - coquille device
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: In this context, an innovative early-stage device was launched in the fall of 2022 at the Coquille unit of the Ville Evrard Public Health Establishment (EPSVE), for children under 30 months with Autism Spectrum Disorder and their families.
  This six-month therapeutic device in day hospital includes:
  * 22 TMF sessions,
  * four two-family observation sessions,
  * three sessions of four unique family sessions,
  * the possibilities of individual targeted intervention in case of need estimated by families and/or caregivers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- coquille device (Other): collaborative family support scheme aimed at improving family functioning and child behaviour
  Interventions: Device: coquille

INTERVENTIONS:
Device: coquille — Modalities: Elaboration of the personalized care project, follow-up parents-child single family, multi-family therapy (MFT).
  Frequency: MFT weekly, bi-familial observation weekly for one month, single-parent child-parent monitoring weekly for five months, MFT father-child bimonthly for six months, three co-parents, three child psychiatric consultations to develop the personalized collaborative care project

SUMMARY:
Collaborative early management of children under 30 months with autism spectrum disorder and their families in an ambulatory child psychiatry unit.

DETAILED DESCRIPTION:
Early intervention in Autism Spectrum Disorder (ASD) is now considered a priority. An approach that targets both child disorders and parental distress, and supports the skills of parents, is desirable. Yet there is no early intervention by the ASD involving parents and targeting both child functioning and parenting skills specifically.

Our objective is to evaluate quantitatively and qualitatively the collaborative family support system for ASD "Coquille". This scheme combines the development of a personalized care project based on parents' priorities, an intensive single-family parent-child follow-up and a group of multi-family therapy , over a total period of 6 months. Our main hypothesis is the significant decrease in behavioral disorders of children, evaluated by CARS, following the Coquille device. Our secondary hypotheses concern the evolution of parental dimensions following the device (sense of coherence, parental skills, parental stress, coping strategies and social support). We assume that these dimensions will change as a result of the scheme, and that they will be maintained in the medium term, six months after Coquille. A semi-structured interview will qualitatively explore the dimensions related to family resources, before and after the follow-up and in the medium term. This will also allow the mother to collect experience of the device.

ELIGIBILITY:
Inclusion Criteria for the mother and the child:

* Age 18 years and over
* French language spoken and written by the parent
* Free and informed consent form , initialled and signed by the parent
* Child under 30 months of age at time of inclusion, diagnosed with autism spectrum disorder
* Total CARS score greater than or equal to 30
* Free and informed consent form, initialled and signed by legal representatives

Exclusion Criteria for the mother only:

* Any acute, somatic or psychiatric clinical condition of the mother not compatible with therapeutic intervention.
* Current engagement in an interventional research protocol
* Mother under protection of justice, guardianship or enhanced curatorship
* Mother no longer having parental authority

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Childhood Autism Rating, Scale, CARS | It is done before the sign of the consent (T-1),
  CARS works by rating your child's behavior, characteristics, and abilities against the expected developmental growth of a typical child.It is done by your primary healthcare provider, a teacher, or a parent by rating the child's behaviors from 1 to 4. 1 being normal for your child's age, 2 for mildly abnormal, 3 for moderately abnormal, and 4 as severely abnormal. Scores range from 15 to 60 with 30 being the cutoff rate for a diagnosis of mild autism. Scores 30-37 indicate mild to moderate autism, while scores between 38 and 60 are characterized as severe autism.
Childhood Autism Rating, Scale, CARS | Six month after the use of coquille device (T1)
  CARS works by rating your child's behavior, characteristics, and abilities against the expected developmental growth of a typical child.It is done by your primary healthcare provider, a teacher, or a parent by rating the child's behaviors from 1 to 4. 1 being normal for your child's age, 2 for mildly abnormal, 3 for moderately abnormal, and 4 as severely abnormal. Scores range from 15 to 60 with 30 being the cutoff rate for a diagnosis of mild autism. Scores 30-37 indicate mild to moderate autism, while scores between 38 and 60 are characterized as severe autism.
Childhood Autism Rating, Scale, CARS | Six month after the follow up (T2)
  CARS works by rating your child's behavior, characteristics, and abilities against the expected developmental growth of a typical child.It is done by your primary healthcare provider, a teacher, or a parent by rating the child's behaviors from 1 to 4. 1 being normal for your child's age, 2 for mildly abnormal, 3 for moderately abnormal, and 4 as severely abnormal. Scores range from 15 to 60 with 30 being the cutoff rate for a diagnosis of mild autism. Scores 30-37 indicate mild to moderate autism, while scores between 38 and 60 are characterized as severe autism.
Sociodemographic and lifestyle | Immediately after the sign of the consent (T0)
  The socio-demographic questionnaire contains 4 items:
  Socio-demographic criteria (gender, date of birth, level of education, marital status and number of children), diet, screen, and sleep.
Sociodemographic and lifestyle | Six month after the use of coquille device (T1)
  The socio-demographic questionnaire contains 4 items:
  Socio-demographic criteria (gender, date of birth, level of education, marital status and number of children), diet, screen, and sleep.
Sociodemographic and lifestyle | Six month after the follow up (T2)
  The socio-demographic questionnaire contains 4 items:
  Socio-demographic criteria (gender, date of birth, level of education, marital status and number of children), diet, screen, and sleep.
Parental Stress Scale | Immediately after the sign of the consent (T0)
  The Parental Stress Scale (PSS) was created in 1995 to measure stress unique to parenting and captures both the joys and demands of parenting. Each following sentences describe feelings and perceptions that relate to the experience of being a parent. The PSS is brief and can be completed in less than 10 minutes. It is an 18-item self-report measure in which parents respond to statements about their typical relationship with their child. The possible range of the PSS is 18 (low stress) to 90 (high stress).
  Respondents indicate how much they agree or disagree to each of the 18 statements. Responses are scored as follows:Strongly disagree = 1,Disagree = 2, Undecided = 3, Agree = 4, Strongly agree = 5
Parental Stress Scale | Six month after the use of coquille device (T1)
  The Parental Stress Scale (PSS) was created in 1995 to measure stress unique to parenting and captures both the joys and demands of parenting. Each following sentences describe feelings and perceptions that relate to the experience of being a parent. The PSS is brief and can be completed in less than 10 minutes. It is an 18-item self-report measure in which parents respond to statements about their typical relationship with their child. The possible range of the PSS is 18 (low stress) to 90 (high stress).
  Respondents indicate how much they agree or disagree to each of the 18 statements. Responses are scored as follows:Strongly disagree = 1,Disagree = 2, Undecided = 3, Agree = 4, Strongly agree = 5
Parental Stress Scale | Six month after the follow up (T2)
  The Parental Stress Scale (PSS) was created in 1995 to measure stress unique to parenting and captures both the joys and demands of parenting. Each following sentences describe feelings and perceptions that relate to the experience of being a parent. The PSS is brief and can be completed in less than 10 minutes. It is an 18-item self-report measure in which parents respond to statements about their typical relationship with their child. The possible range of the PSS is 18 (low stress) to 90 (high stress).
  Respondents indicate how much they agree or disagree to each of the 18 statements. Responses are scored as follows:Strongly disagree = 1,Disagree = 2, Undecided = 3, Agree = 4, Strongly agree = 5
Ways of Coping Checklist | Immediately after the sign of the consent (T0)
  The Ways of Coping Checklist (WCCL; Folkman & Lazarus, 1980) is a checklist of 68 items describing a broad range of behavioral and cognitive coping strategies that an individ- ual might use in a specific stressful episode.They include items from the domains of defensive coping (e.g., avoidance, intellectualization, isolation, suppression), information-seeking, problem- solving, palliation, inhibition of action, direct action, and magical thinking. The checklist is binary, yes or no, and is always answered with a specific stressful event in mind. The items on the WCCL were classified into two categories: problem- focused and emotion-focused.
Ways of Coping Checklist | Six month after the use of coquille device (T1)
  The Ways of Coping Checklist (WCCL; Folkman & Lazarus, 1980) is a checklist of 68 items describing a broad range of behavioral and cognitive coping strategies that an individ- ual might use in a specific stressful episode.They include items from the domains of defensive coping (e.g., avoidance, intellectualization, isolation, suppression), information-seeking, problem- solving, palliation, inhibition of action, direct action, and magical thinking. The checklist is binary, yes or no, and is always answered with a specific stressful event in mind. The items on the WCCL were classified into two categories: problem- focused and emotion-focused.
Ways of Coping Checklist | Six month after the follow up (T2)
  The Ways of Coping Checklist (WCCL; Folkman & Lazarus, 1980) is a checklist of 68 items describing a broad range of behavioral and cognitive coping strategies that an individ- ual might use in a specific stressful episode.They include items from the domains of defensive coping (e.g., avoidance, intellectualization, isolation, suppression), information-seeking, problem- solving, palliation, inhibition of action, direct action, and magical thinking. The checklist is binary, yes or no, and is always answered with a specific stressful event in mind. The items on the WCCL were classified into two categories: problem- focused and emotion-focused.
sense of coherence scale | Immediately after the sign of the consent (T0)
  The Sense of Coherence (SOC) scale evaluates how people perceive life and identifies how they use their resources of resistance to maintain and develop their health.This scale is written by Antonovsky in 1987. There is 13 items. For eachs items, you have to choose between Never, rarely, often, frequently and always.
sense of coherence scale | Six month after the use of coquille device (T1)
  The Sense of Coherence (SOC) scale evaluates how people perceive life and identifies how they use their resources of resistance to maintain and develop their health.This scale is written by Antonovsky in 1987. There is 13 items. For eachs items, you have to choose between Never, rarely, often, frequently and always.
sense of coherence scale | Six month after the follow up (T2)
  The Sense of Coherence (SOC) scale evaluates how people perceive life and identifies how they use their resources of resistance to maintain and develop their health.This scale is written by Antonovsky in 1987. There is 13 items. For eachs items, you have to choose between Never, rarely, often, frequently and always.
Parent Sense of Competency Scale (PSOC) | Immediately after the sign of the consent (T0)
  The Parenting Sense of Competency Scale (PSOC) was developed by Gibaud-Wallston as part of her PhD dissertation and presented at the American Psychological Association by Gibaud-Wallston and Wandersman in 1978. The PSOC is a 17 item scale, with 2 subscales. Each item is rated on a 6 point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree".
  Nine (9) items (#s 2, 3, 4, 5, 8, 9, 12, 14, and 16) on the PSOC are reverse coded.
Parent Sense of Competency Scale (PSOC) | Six month after the use of coquille device (T1)
  The Parenting Sense of Competency Scale (PSOC) was developed by Gibaud-Wallston as part of her PhD dissertation and presented at the American Psychological Association by Gibaud-Wallston and Wandersman in 1978. The PSOC is a 17 item scale, with 2 subscales. Each item is rated on a 6 point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree".
  Nine (9) items (#s 2, 3, 4, 5, 8, 9, 12, 14, and 16) on the PSOC are reverse coded.
Parent Sense of Competency Scale (PSOC) | Six month after the follow up (T2)
  The Parenting Sense of Competency Scale (PSOC) was developed by Gibaud-Wallston as part of her PhD dissertation and presented at the American Psychological Association by Gibaud-Wallston and Wandersman in 1978. The PSOC is a 17 item scale, with 2 subscales. Each item is rated on a 6 point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree".
  Nine (9) items (#s 2, 3, 4, 5, 8, 9, 12, 14, and 16) on the PSOC are reverse coded.
Multidimensional Scale of Perceived Social Support (MSPSS) | Immediately after the sign of the consent (T0)
  The Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item questionnaire to identify an individual's perceived level of social support with family, friends, and significant others.
Multidimensional Scale of Perceived Social Support (MSPSS) | Six month after the use of coquille device (T1)
  The Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item questionnaire to identify an individual's perceived level of social support with family, friends, and significant others.
Multidimensional Scale of Perceived Social Support (MSPSS) | Six month after the follow up (T2)
  The Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item questionnaire to identify an individual's perceived level of social support with family, friends, and significant others.
The Marlowe-Crowne Social Desirability Scale (MC-SDS) | Immediately after the sign of the consent (T0)
  The social desirability scale is a 33-items self-report questionnaire that assesses whether or not respondents are concerned with social approval. The scale was created by Douglas P. Crowne and David Marlowe in 1960 in an effort to measure social desirability bias, which is considered one of the most common biases affecting survey research.A high number of socially desirable responses might indicate that the respondent is generally concerned with social approval and conforming to societal conventions, while a low score might indicate that the respondent is less concerned with such things and is more willing to answer survey questions truthfully and representing themselves accurately.
The Marlowe-Crowne Social Desirability Scale (MC-SDS) | Six month after the use of coquille device (T1)
  The social desirability scale is a 33-items self-report questionnaire that assesses whether or not respondents are concerned with social approval. The scale was created by Douglas P. Crowne and David Marlowe in 1960 in an effort to measure social desirability bias, which is considered one of the most common biases affecting survey research.A high number of socially desirable responses might indicate that the respondent is generally concerned with social approval and conforming to societal conventions, while a low score might indicate that the respondent is less concerned with such things and is more willing to answer survey questions truthfully and representing themselves accurately.
The Marlowe-Crowne Social Desirability Scale (MC-SDS) | Six month after the follow up (T2)
  The social desirability scale is a 33-items self-report questionnaire that assesses whether or not respondents are concerned with social approval. The scale was created by Douglas P. Crowne and David Marlowe in 1960 in an effort to measure social desirability bias, which is considered one of the most common biases affecting survey research.A high number of socially desirable responses might indicate that the respondent is generally concerned with social approval and conforming to societal conventions, while a low score might indicate that the respondent is less concerned with such things and is more willing to answer survey questions truthfully and representing themselves accurately.
Aberrant Behavior Checklist | Immediately after the sign of the consent (T0)
  The Aberrant Behavior Checklist consists of 58 questions across 5 different domains: (a) irritability, (b) social withdrawal, (c) stereotypic behavior, (d) hyperactivity/noncompliance, and (e) inappropriate speech. The rater has to answer each of the 58 questions using a 4-point Likert scale. A score of a "0" means the behavior is not a problem, a score of a "1" means slight problem, a score of a "2" means a serious problem, and a "3" means a severe problem.
Aberrant Behavior Checklist | Six month after the use of coquille device (T1)
  The Aberrant Behavior Checklist consists of 58 questions across 5 different domains: (a) irritability, (b) social withdrawal, (c) stereotypic behavior, (d) hyperactivity/noncompliance, and (e) inappropriate speech. The rater has to answer each of the 58 questions using a 4-point Likert scale. A score of a "0" means the behavior is not a problem, a score of a "1" means slight problem, a score of a "2" means a serious problem, and a "3" means a severe problem.
Aberrant Behavior Checklist | Six month after the follow up (T2)
  The Aberrant Behavior Checklist consists of 58 questions across 5 different domains: (a) irritability, (b) social withdrawal, (c) stereotypic behavior, (d) hyperactivity/noncompliance, and (e) inappropriate speech. The rater has to answer each of the 58 questions using a 4-point Likert scale. A score of a "0" means the behavior is not a problem, a score of a "1" means slight problem, a score of a "2" means a serious problem, and a "3" means a severe problem.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre LECARPENTIER, MBBS, Principal Investigator — EPS VILLE EVRARD
Locations (1):
- Eps Ville Evrard, Neuilly-sur-Marne, France

IPD SHARING:
Plan to Share IPD: No